CLINICAL TRIAL: NCT01817387
Title: Developing an Intervention Strategy to Enhance Motivation in Recent Onset Schizophrenia
Brief Title: Enhancing Motivation in Recent Onset Schizophrenia
Acronym: PRIME
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to participants not completing the cognitive training requirement.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: NIMHK23SCH
Record Dates: First submitted 2013-03-13; First posted 2013-03-25 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PRIME + CT (Experimental): 4 months use of PRIME mobile application on mobile device and 30 hours of cognitive training
  Interventions: Behavioral: PRIME; Behavioral: Cognitive Training
- Daily Goals + CT (Experimental): 4 months use of Daily Goals mobile application on mobile device and 30 hours of cognitive training
  Interventions: Behavioral: Cognitive Training

INTERVENTIONS:
Behavioral: PRIME — Mobile application designed to improve psychosocial functioning and motivational deficits
  Arms: PRIME + CT
Behavioral: Cognitive Training — Auditory processing, verbal learning, memory, processing speed, and social cognition

SUMMARY:
This project will result in the development of a personalized intervention strategy to improve motivation for treatment engagement and functional outcomes in individuals with a recent onset of schizophrenia. Motivational impairment is arguably the single most important factor that determines a patient's ability to engage in and adhere to effective treatment. In our study, sixty participants will be enrolled in a randomized controlled trial comparing the feasibility and tolerability of two types of motivational interventions (Daily Goals or PRIME), and a neuroplasticity-based cognitive training program. Participants are randomized to either receive Daily Goals or PRIME for 8 weeks, after which, both conditions will also receive an 8-week course of cognitive training delivered via iPads. Participants will undergo pre/post-testing and a 6-month follow-up to determine feasibility and efficacy of the interventions. By enhancing motivation, schizophrenia patients would be able to engage more fully with treatment and develop full and productive lives. This study may also pave the way forward for other health conditions in which motivational impairments impede health outcomes.

All assessments will be conducted at the University of California, San Francisco; however, we offer some assessments to be done remotely.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia, schizoaffective, or schizophreniform disorder.
* Onset of diagnosis within 5 years.
* 14-30 years old.
* Clinically stable (outpatient status for 1 month and stable dose of medication for 1 month).
* Good general health

Exclusion Criteria:

* Substance dependence within the past 12 months,
* Current substance abuse,
* No history of neurological disorder

Ages: 14 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2014-07; Primary Completion 2018-03-20 (Actual); Study Completion 2018-03-20 (Actual)

PRIMARY OUTCOMES:
Psychosocial functioning | past 30 days
  Work status, work performance, social status, social performance, health status, health performance

CONTACTS AND LOCATIONS:
Overall Officials: Danielle A Schlosser, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No